CLINICAL TRIAL: NCT05613361
Title: The Effect of Curcumin Against Colistin-induced Nephrotoxicity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Hammad, Principal Investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: curcumin in nephrotoxicity
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Acute Kidney Injury; Drug-Induced Nephropathy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Colistin; Curcumin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): patients in this group will receive loading dose of colistin intravenously of 9 MIU followed by maintenance doses of 4.5 MIU given every 12 hours.
  Interventions: Drug: Colistin
- Group 2 (Active Comparator): patients in this group will receive loading dose of colistin intravenously of 9 MIU followed by maintenance doses of 4.5 MIU given every 12 hours and curcumin will be administered as orally or through nasogastric tube at a dose of 2 capsules every 6 hours (1 gm/6 hour)
  Interventions: Drug: Colistin; Drug: Curcumin

INTERVENTIONS:
Drug: Colistin — added for infection with multi drug resistant bacteria
Drug: Curcumin — added for the possible nephroprotective effect
  Arms: Group 2

SUMMARY:
The goal of this study is to investigate the possible nephroprotective effect of curcumin in critically ill patients receiving colistin.

DETAILED DESCRIPTION:
The study will investigate the possible nephroprotective effect of curcumin when added to patients infected by MDR Gram-negative bacteria and require intravenous colistin therapy, curcumin will be given concurrently with colistin and discontinued at the same time as Colistin.

ELIGIBILITY:
Inclusion Criteria:

* All critically ill adult patients (18-65 years old) who are infected by MDR Gram-negative bacteria and require intravenous colistin therapy

Exclusion Criteria:

* Patients receiving intravenous colistin therapy for < 72 hours.
* Patients receiving renal replacement therapy (RRT).
* Patients with diseases that may contribute to renal impairment such as systemic lupus erythematosus, acute myocardial infarction, cancer, HIV infection, glucose-6-phosphate-dehydrogenase deficiency, or urinary tract stone.
* Pregnancy or breastfeeding.
* Known allergy to the study medications.
* Patients with chronic kidney diseases (creatinine clearance < 60 mg/dL).
* Elevated total liver enzymes (AST, and ALT) three times above the upper limit of normal.
* Patients with acute decompensated heart failure signs and symptoms requiring intravenous loop diuretics and/or intravenous inotropes and/or ACE inhibitors.
* Uncontrolled diabetes (Glycosylated hemoglobin (Hb A1C) >8%).
* Hypotensive patients defined as decrease in blood pressure less than 90/60 mm Hg.
* Recent use of vitamins with antioxidant properties such as beta carotene, vitamin E, vitamin C, selenium, or N-acetylcysteine or any other medications known to have nephroprotective activities.
* Patients receiving other nephrotoxic drugs at enrollment (e.g., aminoglycosides, vancomycin, or amphotericin B) or administration of contrast medium within 7 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of acute kidney injury | Baseline to hospital discharge, an average of 14 days.
  colistin induced nephrotoxicity (CIN) is defined as increase of serum creatinine by 0.3 mg/dL 48 hours after colistin administration

SECONDARY OUTCOMES:
The incidence of acute tubular necrosis (ATN) | Baseline to hospital discharge, an average of 14 days.
  will be evaluated by fractional excreted sodium (FENa)
The difference between the levels of urinary NGAL | Baseline to hospital discharge, an average of 14 days.
Mortality rate | Baseline to 30 days post discharge
Total length of ICU and hospital stays. | Baseline to hospital discharge, an average of 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmeen A. Sabry, Principal Investigator — Professor of Clinical Pharmacy Faculty of Pharmacy Cairo University; Maggie M. Abbassi, Principal Investigator — Professor of Clinical Pharmacy Faculty of Pharmacy Cairo University; Rania El-Husseiny, Principal Investigator — Professor of Critical Care Medicine, Faculty of Medicine Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes